CLINICAL TRIAL: NCT05245448
Title: Comparing the Efficacy of Tetrandrine Combined With Methotrexate and Methotrexate Alone in the Treatment of Rheumatoid arthritis---a Randomized, Double-blinded, Placebo-controlled, Multicenter Study
Brief Title: Tetrandrine in the Treatment of Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-Z-40
Record Dates: First submitted 2022-01-22; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; tetrandrine
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tetrandrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tetrandrine (Experimental): tetrandrine administered 40milligram (mg) orally thrice daily through Week 24.
  Interventions: Drug: Tetrandrine
- placebo (Placebo Comparator): Placebo administered orally thrice daily through Week 12. Starting at Week 12, participants were given tetrandrine 40 milligram (mg) orally thrice daily through Week 24.
  Interventions: Drug: Tetrandrine; Drug: Placebo

INTERVENTIONS:
Drug: Tetrandrine — Administered orally
Drug: Placebo — Administered orally
  Arms: placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of tetrandrine, compared with placebo in 12 week or 24 week in RA patients with inadequate response to methotrexate.

DETAILED DESCRIPTION:
The investigators designed a randomized, double-blinded, placebo-controlled, multicenter study. Adults with active rheumatoid arthritis and inadequate response to methotrexate will be enrolled, meeting the 1987 revised American College of Rheumatology (ACR) or 2010 ACR & European alliance of associations for rheumatology (EULAR) classification criteria. Two hundred forty patients at 18 to 65 years of age will be enrolled in the study, and be randomly assigned (in a 1:1 ratio) to one of the two arms (group1: tetrandrine 40mg tid for 24 weeks or group 2: placebo two tablets tid for 12 weeks, and then 40mg tid for 12 weeks). Follow-up visits will occur on weeks 4, 12 and 24. The end points were 20% improvement in American College of Rheumatology criteria (ACR20) in 12 week.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old.
* fulfilled the 1987 revised American College of Rheumatology (ACR) or 2010 ACR/EULAR classification criteria for RA.
* DAS28-ESR>3.2.
* MTX 7.5-20mg/w for at least 12 weeks before screening and keep stable doses for at least 4 weeks.
* Prednisone (≤10mg/d) or equivalent dose is allowed. However, the dose should be stable for at least 4 weeks before screening and should not increase during follow-up. If glucocorticoids are not used before screening, short- and intermediate-acting glucocorticoids should have been stopped at least 1 week and long-acting glucocorticoids should have been stopped at least 2 weeks.

Exclusion Criteria:

* Allergic to the drugs involved in the study, or allergic to more than two kinds of food or drugs or pollen.
* Meets the ACR 1991 Revised Criteria for the Classification of Global Functional Status in RA Class IV in the Screening Phase.
* Any history or complication of other autoimmune diseases other than Sjogren's syndrome or Hashimoto Thyroiditis.
* Current active infections.
* Tested positive for any of the following in the Screening Phase: HIV, hepatitis B virus surface antigen (HBs antigen), hepatitis B virus surface antibody (HBs antibody), hepatitis C virus antibody (HCV antibody), or history of AIDs.
* Females of childbearing or breastfeeding.
* Presence of any unstable cardiovascular disease (including congestive heart failure with NYHA class III or IV, unstable angina pectoris, history of myocardial infarction within one year), and the presence of conditions that can lead to QTc prolongation or arrhythmia.
* Presence of progressive, uncontrolled cerebrovascular disease, hematopoietic, endocrine (including diabetes), respiratory (including interstitial pneumonia and pulmonary fibrosis) and other serious diseases and psychiatric diseases, or the investigator believes that participation in the study would place the subject at unacceptable risk.
* History of malignancy.
* Laboratory tests during screening：i. WBC<3.5×109/L，PLT<90×109/L， Hb<90g/L; ii. ALT or AST>1.5ULN; iii. Scr>ULN.
* Use of iguratimod or disease-modifying antirheumatic drugs (DMARDs) other than MTX (such as leflunomide, sulfasalazine, hydroxychloroquine, D- penicillamine, azathioprine, cyclosporine, cyclophosphamide, Tripterygium, etc.) within 4 weeks before enrollment.
* Use of traditional Chinese medicines for rheumatoid arthritis within 4 weeks before enrollment.
* Use of b/tsDMARDs within 12 weeks.
* History of alcohol and drug abuse.
* The investigator or subinvestigator would compromise the participant's ability to safely complete the study.
* Participate in other clinical trial within 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-02-22 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving American College of Rheumatology (ACR) 20 | week 12
  The ACR20 was achieved if there was at least a 20% improvement from baseline in swollen joint count 66 (SJC66) and tender joint count 68 (TJC68) and 3 or more of the 5 following assessments: participant's assessment of pain, GH, physician's global assessment of disease activity, participant's assessment of physical function and CRP.

SECONDARY OUTCOMES:
Proportion of Participants Achieving American College of Rheumatology (ACR) 20 | week 4 and week 24
  The ACR20 was achieved if there was at least a 20% improvement from baseline in swollen joint count 66 (SJC66) and tender joint count 68 (TJC68) and 3 or more of the 5 following assessments: participant's assessment of pain, GH, physician's global assessment of disease activity, participant's assessment of physical function and CRP.
Proportion of Participants Achieving American College of Rheumatology (ACR) 50 and ACR70 | week 12 and week 24
  The ACR50 or ACR70 was achieved if there was at least a 50% or 70% improvement from baseline in swollen joint count 66 (SJC66) and tender joint count 68 (TJC68) and 3 or more of the 5 following assessments: participant's assessment of pain, GH, physician's global assessment of disease activity, participant's assessment of physical function and CRP.
Rates of European League Against Rheumatism (EULAR) Response Using DAS28-CRP | week 12 and week 24
  The Disease Activity Score Based on 28-joints Count based EULAR response criteria was used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28-CRP <=3.2; moderate responders: change from baseline >1.2 with DAS28-CRP >3.2 to <=5.1 or change from baseline >0.6 to <=1.2 with DAS28-CRP <=5.1; non-responders: change from baseline <=0.6 or change from baseline >0.6 and <=1.2 with DAS28-CRP >5.1.
Change From Baseline in Disease Activity Score 28 (DAS28)-CRP | Baseline, week 4, week 12 and week 24
  The DAS28 index was a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, participant global assessment of disease activity score, and CRP value. A positive change in score indicates worsening, and a negative change indicates improvement.
Change From Baseline in Pain VAS Score | Baseline, week 4, week 12 and week 24
  Pain assessments are reported by placing a mark on a 100 millimeter horizontal VAS. The scale ranged from 0-100 mm, where 0 indicated no pain and 100 represented maximum pain).
Change From Baseline in C-reactive Protein (CRP) Values | Baseline, week 4, week 12 and week 24
  CRP (milligrams per deciliter) are blood tests.
Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) | Baseline, week 4, week 12 and week 24
  The degree of disability was self-evaluated by the participant using the HAQ-DI. The minimum value is 0, and the maximum values is 3. Higher scores mean a worse outcome.
Change From Baseline to Week 24 in OMERACT RAMRIS Wrist and MCP Bone Marrow Edema. | Baseline and week 12
  Bone edema was assessed at 25 locations: 15 in 1 wrist and 10 in attached hand. Bone edema was defined as a lesion within the trabecular bone, with ill-defined margins and signal characteristics consistent with increased water content. Each bone was scored separately; the scale was 0-3 based on the proportion of bone with edema, as follows 0: no edema; 1: 1-33% of bone edematous; 2: 34-66% of bone edematous; 3: 67-100%. OMERACT RAMRIS total bone edema score for hands/wrists was sum of the individual scores for each location. The maximum score per hand/wrist was 75 (range 0-75). Increasing score indicates greater severity.
Change From Baseline in immune cells | Baseline, week 12 and week 24
  The percentages of immune cells, such as T/B/NK and Th subsets will be detected.
Change From Baseline in Simplified Disease Activity Index (SDAI) Score | Baseline, week 4, week 12 and week 24
  The SDAI was calculated from tender joint counts of 28, swollen joint counts of 28, participant's global assessment of disease activity, physician global assessment of disease activity score, and CRP value. A positive change in score indicates worsening, and a negative change indicates improvement.
Change From Baseline in Clinical Disease Activity Index (CDAI) Score | Baseline, week 4, week 12 and week 24
  The CDAI was calculated from tender joint counts of 28, swollen joint counts of 28, participant's global assessment of disease activity, physician global assessment of disease activity score. A positive change in score indicates worsening, and a negative change indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Department of Rheumatology and Immunology, Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China